CLINICAL TRIAL: NCT04530474
Title: Outpatient Use of Ivermectin in COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: WHO report
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1285242
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: IVERMECTIN; COVID
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Experimental): Single dose of 0.15-2 mg/kg/dose to a maximum of 12 mg
  Interventions: Drug: Ivermectin Pill
- Placebo (Placebo Comparator): Single dose of 2-4 placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin Pill — Ivermecin as a one-time dose
  Arms: Ivermectin
Drug: Placebo — Inactive medication as a one time dose
  Arms: Placebo

SUMMARY:
Covid 19, a novel coronavirus, causes infection that, while mild to moderate in many people, can lead to severe disease in a significant portion. Currently, it is expected that the majority, 81%, of patients with COVID-19 will have mild to moderate disease, with 14% having more severe disease (2). There exists a number of candidate drugs that may inhibit SARS-CoV-2 infection or progression of disease. Simple, safe and low-cost strategies that may be the best solution to inhibit infection and limit transmission and spread of infection.

Ivermectin is a drug initially synthesized and used as an anthelmintic. It has been found to have activity against several RNA viruses such as the SARS-CoV-2 by mechanisms that inhibit importin α/β-mediated nuclear transport that may prevent viral proteins from entering the nucleus to alter host cell function. A recent in vitro study showed that a single dose of ivermectin could kill COVID-19 in vitro within 48 hours. A recent multi-continent retrospective study of 1,400 patients demonstrated an association of ivermectin use with lower in-hospital mortality 1.4% versus 8.5%. Given these findings and its safety profile, cost and ease of administration, Ivermectin warrants study as a potential treatment to prevent progression of COVID 19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms highly suspicious for COVID-19.
2. Age at least 18 years
3. Negative pregnancy test for women of child bearing age
4. Able to consent to participate in the study.

Exclusion Criteria:

1. Known history of Ivermectin allergy
2. Hypersensitivity to any component of Stromectol®
3. COVID-19 Pneumonia identified by chest X-ray or high resolution CT scan
4. Fever or cough present for more than 7 days
5. Positive IgG against SARS-CoV-2 by rapid test if available on baseline screening.
6. The following co-morbidities (or any other disease that, in the opinion of the investigators, might interfere with the study:

   1. Immunosuppression
   2. HIV
   3. Acute or chronic renal failure
   4. Current neoplasm
7. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal within the prior 6 months if available OR clinical evidence of liver failure with jaundice, ascites, encephalopathy.
8. Current use of CYP 3A4 or P-gp inhibitor drugs such as quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir or cobicistat. Use of critical CYP3A4 substrate drugs such as warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | 28 days
  Clinical Improvement as measured by the inFLUenza Patient-Reported Outcome (FLU-PRO)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No